CLINICAL TRIAL: NCT00512941
Title: Laboratory Profile of Hepatitis B and C in Users of a Reference Service
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Sergio Muller, Faculdade de Medicina de Botucatu - Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-15
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Hepatitis, Viral, Non-A, Non-B, Parenterally-Transmitted; Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- 1: HBV: Carrier
- 2: HBV: cure
- 3: HBV: isolate anti-HBc
- 4: HBV: vaccinated
- 5: HCV: anti-HCV positive test
- 6: HBV/HCV co-infection
- 7: Susceptible individuals

SUMMARY:
Chronic hepatitis by the B virus (HBV) and/or by the C virus (HCV) is a major public-health problem since it presents a long phase of clinical latency which makes its early diagnosis difficult and results in the development of a large number of cases to complications such as cirrhosis, hepatic insufficiency and hepatocarcinoma. In Brazil, it is estimated that the number of HBV is two million, of which 72 thousand have been reported. As regards HCV, the ratio is one of three million estimated cases to 52 thousand reports. Learning about the serological profile of the users of a viral hepatitis reference service is fundamental for the planning of diagnostic and caregiving actions; therefore, it is the objective of this study.

DETAILED DESCRIPTION:
Chronic hepatitis by virus B (HVB) and/or by virus C (HVC) is a major public-health problem since it presents a long phase of clinical latency which makes its early diagnosis difficult and results in the development of a large number of cases to complications such as cirrhosis, hepatic insufficiency and hepatocarcinoma. In Brazil, it is estimated that the number of HVB patients is two million, but only 72 thousand have been reported. As regards HVC, the ratio is three million estimated cases to 52 thousand reports. Learning about the serological profile of the users of a viral hepatitis reference service is essential for the planning of diagnostic and therapeutic actions; therefore, it is the objective of this study.

Five hundred and thirty-one HVB and HVC serological profiles of the patients referred to SAE/HD within a period of 18 months (January 2006 to June 2007) were studied by means of retrospective analysis. The patients were classified as: a) HBV: carrier, cure, isolated anti-HBc and vaccinated; b) HVC: reagent anti-HVC; c) HBV/HVC co-infection: AgHBs and reagent anti-HVC; and d) Susceptible: non-reagent serology.

As regards HBV, the following were found from the total number of patients: carriers, 12.6%; cure, 18.9%; isolated anti-HBc, 9.0% and vaccinated, 6.2%. The patients with reagent anti-HVC comprised 31.3% of the total number of individuals. HBV/HCV co-infection was 0.6%. Susceptible individuals comprised 20.5%.

It was concluded that approximately 45% of the referred patients carried chronic infection by B and/or C virus, a condition which requires additional investigation and, in many instances, specific treatment. Strategies for early diagnosis are essential in order to prevent the intrinsic complications of such condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with laboratory tests positive for hepatitis B and/or C

Exclusion Criteria:

* No laboratory tests available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with laboratory tests positive for hepatitis B and/or C
Sampling Method: Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2007-06; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre N Barbosa, MD, MSc, Principal Investigator — SAE e Hospital Dia de Aids
Locations (2):
- Brazil (2):
  - SAE e Hospital Dia de Aids, Botucatu, São Paulo
  - SAE e Hospital Dia, Botucatu, São Paulo